CLINICAL TRIAL: NCT05675254
Title: The Prevalence and Risk Factors of Coagulopathy in Pediatric Patients Undergoing Surgery for Epilepsy
Brief Title: The Prevalence and Risk Factors of Coagulopathy in Pediatric Epilepsy Surgery Patients
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: No. 2022-355
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy in Children; Coagulation and Hemorrhagic Disorders; Epilepsy; Seizure; Antiepileptic Adverse Reaction
Keywords: Pediatric; Epilepsy; Surgery; Coagulation Function; Anti-seizure Medications
MeSH Terms: conditions — Thrombosis; Hemorrhagic Disorders; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EP with ASMs: Epilepsy patients who administered Anti-seizure Medications(ASMs)
- EP without ASMs: Epilepsy patients who were not administered ASMs
- No EP: Non-epileptic children and had never taken any ASMs

SUMMARY:
The hematologic consequences of novel Anti-seizure medications (ASMs) are rarely reported.

Whether coagulation dysfunctions increase the risk of peri-operative bleeding remains controversial.

The research is performed to investigated the incidence and risk factors of preoperative coagulation dysfunction in children undergoing surgery for epilepsy and their impact on surgery.

DETAILED DESCRIPTION:
Epilepsy is a common disease of the nervous system with severe consequences. Epidemiological surveys have shown that the prevalence of epilepsy in China is approximately 0.4-0.7%, comprising 7-10 million patients with epilepsy, most of whom are children. Although most symptoms of epilepsy can be controlled with the use of anti-seizure medications (ASMs), there are still a few patients who cannot achieve satisfactory seizure control with such medications or cannot tolerate their side effects, thus requiring surgical treatment. Surgical treatment of epilepsy has been recognized as a valuable treatment option for carefully selected patients to achieve better seizure control and quality of life. Compared to adults, children with epilepsy with indications for surgery usually have a better prognosis after surgical treatment. Many children undergoing surgery for epilepsy have a long history of using ASMs. Moreover, ASM therapy usually consists of multiple varieties of drugs, thereby bringing significant attention to the side effects of ASMs, especially those that may be relevant in the perioperative surgical setting.

ASMs have been associated with multiple adverse effects on platelets and the coagulation system. Valproic acid (VPA), one of the most commonly used traditional ASM, has been reported to cause multiple hematologic abnormalities, including thrombocytopenia, platelet aggregation dysfunction, fibrinogen (FBG) depletion, bone marrow suppression, decreased factor XIII, and acquired von Willebrand disease. However, the wide use of novel ASMs in recent decades has led to decreased reports of adverse events. The hematologic consequences of these novel ASMs or combined therapies are rarely reported. Few studies have suggested that levetiracetam (LEV) does not cause clinically significant or relevant hematological disorders.

Such reported side effects may be more significant in pediatric patients with epilepsy due to individual differences in age, weight, and pharmacokinetic action of the body on the drugs. The incidence of coagulopathies has been reported to be higher in children than in adults, especially hypofibrinogenemia. Nevertheless, whether these coagulation dysfunctions increase the risk of peri-operative bleeding remains controversial. Most investigators suggest that ASMs, including VPA, are not associated with surgery-related blood loss or transfusion requirements. However, a few studies have suggested that considering the extra risk of peri-operative bleeding, VPA should be discontinued before surgery.

This retrospective analysis of 390 children with epilepsy systematically investigated the incidence and risk factors of preoperative coagulation dysfunction in children undergoing surgery for epilepsy and their impact on surgery, with the objective to provide detailed and valuable clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Age<18 years
* A discharge diagnosis of "epilepsy" according to the International Classification of Diseases (ICD-10)
* Received surgical treatment for epilepsy during the hospitalization
* Hospitalized between January 2015 and December 2021 at the Neurosurgery Department of Children's Hospital of Fudan University
* Non-epileptic children who underwent non-epilepsy neurological surgery by the same surgeon and were admitted at the same period for control

Exclusion Criteria:

* The clinical information or laboratory examinations were incomplete
* Had concomitant diseases affecting coagulation or liver function
* Patients or parents refused to be enrolled

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population were children who were hospitalized between January 2015 and December 2021 at the Neurosurgery Department of Children's Hospital of Fudan University, including non-epileptic children who underwent non-epilepsy neurological surgery by the same surgeon and were admitted at the same period for control.
  * 319 patients with epilepsy who administered Anti-seizure Medications (ASMs);
  * 71 patients with epilepsy who were not administered ASMs;
  * 104 non-epileptic children who underwent neurosurgical operations and had never taken any ASMs.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Factors related to coagulation function | From hospitalization to surgery, an average of 3 days
  The following clinical data were collected: sex, age, weight, epilepsy course, and anti-seizure therapy. The initial laboratory data after admission included platelet count (PLT), prothrombin time (PT), activated partial thromboplastin time (APTT), FBG, alanine aminotransferase (ALT), and aspartate aminotransferase (AST).
  We also collected data on non-epileptic children who underwent non-epilepsy neurological surgery and were admitted at the same period from the Hospital Information System (HIS) as a control cohort.
  Multivariate logistic regression analysis was performed to identify independent determinants of coagulation dysfunction. Possible relevant variables were filtered out using univariate logistic regression and further included as covariates for the multivariate logistic regression.

SECONDARY OUTCOMES:
Proportion of coagulation dysfunction between groups | From hospitalization to surgery, an average of 3 days
  Proportion of cases with or without coagulation dysfunction in epileptic children with ASMs, epileptic children without ASMs, and non-epileptic children.
Variables affecting coagulation function | From hospitalization to surgery, an average of 3 days
  Univariate analysis and logistic regression identified the risk factors for coagulopathy in paediatric patients undergoing epilepsy surgery.
Affected laboratory index | From hospitalization to surgery, an average of 3 days
  Laboratory index affected by the independent determinants of coagulation dysfunction (PT, APTT, FBG or PLT).
Incidence of transfusion | From surgery to discharge, an average of 7 days
  Whether the independent determinants of coagulation dysfunction increase the incidence of surgical-related transfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
According to the Ethic Board of Children's Hospital of Fudan University, the clinical data of patients could not been shared without permission.

REFERENCES:
- [Derived] Zhu R, Wang Q, Zhou Y, Shi W, Zhang Y, Wang M, Li H, Zhao R. The prevalence and risk factors of coagulopathy in pediatric patients undergoing surgery for epilepsy. J Neurosurg Pediatr. 2023 Aug 18;32(5):527-534. doi: 10.3171/2023.6.PEDS23196. Print 2023 Nov 1. PMID 37728406

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT05675254/Prot_SAP_000.pdf